CLINICAL TRIAL: NCT01535443
Title: Fase 1 Study to Evaluate the Safety and Tolerability of PRO-155 Ophthalmic Solution 0.09% in Healthy Volunteers.
Brief Title: Safety and Tolerability of PRO-155 Ophthalmic Solution 0.09% in Healthy Volunteers.
Acronym: PRO-155
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRON0611V1FI
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Results first posted 2019-07-19 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Inflammation; Cataract
Keywords: PRO-155; Ocular NSAIDs; Safety and tolerability; Ocular Inflammation; Ocular Paint
MeSH Terms: conditions — Inflammation; Cataract | interventions — bromfenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bromfenac (Experimental): Drug: Bromfenac ophthalmic solution 1 drop 4 times per day
  Interventions: Drug: Bromfenac

INTERVENTIONS:
Drug: Bromfenac — Drug: Bromfenac Other names: PRO-155
  Other Names: PROJECT SOPHIA PRO-155

SUMMARY:
Study to evaluate the safety and tolerability of PRO-155 Ophthalmic Solution 0.09 % in healthy volunteers.

DETAILED DESCRIPTION:
A phase I, open label and unicentric clinical trial to evaluate the safety and tolerability of PRO-155 Ophthalmic Solution 0.09 % in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female.
* Age ≥ 18 years old at screening visit

Exclusion Criteria:

* Any ocular or systemic condition.
* Patient with one blind eye.
* Visual acuity of 20/40 in any eye.
* Use of ocular or systemic medications.
* Contraindications or sensitivity to any component of the study treatments.
* Contact lens users.
* Ocular surgery within the past 3 months..
* Women who were not using an effective means of contraception or who were pregnant or nursing.
* Participation in any studies of investigational drugs within 90 days previous to the inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Lizarraga-Corona, MD, Principal Investigator — Unidad Medica "Grupo Pediátrico"; Leopoldo M Baiza-Duran, MD, Study Director — Clinical Research Department. Laboratorios Sophia SA de CV
Locations (1):
- Unidad Medica "Grupo Pediátrico", Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PRO-155 Ophthalmic Solution 0.09 %: PRO-155 Ophthalmic Solution 0.09 % : PRO-155 Ophthalmic Solution 0.09 % applied twice a day during 10 days..
Period: Overall Study
Arm/Group | PRO-155 Ophthalmic Solution 0.09 %
Started | 35
Completed | 32
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Groups:
- PRO-155 Ophthalmic Solution 0.09 %: PRO-155 Ophthalmic Solution 0.09 % : PRO-155 Ophthalmic Solution 0.09 % applied twice to day during 10 days..
Arm/Group | PRO-155 Ophthalmic Solution 0.09 %
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 19
Region of Enrollment [Number; unit: participants]
  Mexico | 35

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: A Snellen chart is an eye chart that can be used to measure visual acuity. consisting of a scale ranging from 20 to 200, where 20 is the best visual capacity and 200 is the worst
Time Frame: 10 days
Population: Per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | PRO-155 Ophthalmic Solution 0.09 %
Number analyzed (Participants) | 34
Number analyzed (eyes) | 68
units on a scale
  right eye | 20.3 (1.2)
  left eye | 20.2 (0.9)
Statistical Analysis 1: Comparison: PRO-155 Ophthalmic Solution 0.09 %; Test type: Other; p = .374, Traza Pillai; The test was performed with degrees of freedom: 2

2. Secondary Outcome: Adverse Events
Description: will be reported the presence of adverse events presented in the study group during the intervention period .
Time Frame: 10 days
Population: Analysis by intention to treat (ITT)
Measure: Number; unit: events
Units Other Than Participants: eyes
Arm/Group | PRO-155 Ophthalmic Solution 0.09 %
Number analyzed (Participants) | 35
Number analyzed (eyes) | 70
events | 1

3. Secondary Outcome: Findings in Posterior Segment
Description: Abnormal bores will be reported when assessing the integrity of the posterior segment, the unit of measure will be number of findings.
Time Frame: 10 days
Measure: Number; unit: abnormal findings
Units Other Than Participants: eyes
Arm/Group | PRO-155 Ophthalmic Solution 0.09 %
Number analyzed (Participants) | 34
Number analyzed (eyes) | 68
abnormal findings
  right eye | 1
  left eye | 1

4. Secondary Outcome: Intraocular Pressure (IOP)
Description: Intraocular pressure (IOP) measurement by applanation tonometry. The unit of measurement will be millimeters of mercury (mmhg) the normal range will be considered 11 to 21 mmhg.
Time Frame: 10 days
Population: Analyze by intention to treat
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmhg)
Arm/Group | PRO-155 Ophthalmic Solution 0.09 %
Number analyzed (Participants) | 35
millimeters of mercury (mmhg)
  right aye | 13.3 (2.1)
  left eye | 13.4 (2)

5. Secondary Outcome: Hyperemia
Description: The red eye will be evaluated by the absence or presence of hyperemia.
Time Frame: 10 days
Population: Intention to treat analysis (ITT)
Measure: Number; unit: eyes
Arm/Group | PRO-155 Ophthalmic Solution 0.09 %
Number analyzed (Participants) | 35
eyes
  right eye | 0
  left eye | 0

6. Secondary Outcome: Burning
Description: Eye ocular burning will be reported according to the following scale: absent, mild, moderate and severe.
Time Frame: 10 days
Population: Intention-to-treat analysis (ITT)
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | PRO-155 Ophthalmic Solution 0.09 %
Number analyzed (Participants) | 35
Number analyzed (eyes) | 70
eyes
  right eye : absent | 34
  right eye : mild | 0
  right eye : moderate | 0
  right eye : severe | 0
  left eye : absent | 33
  left eye : mild | 0
  left eye : moderate | 0
  left eye : severe | 1

7. Secondary Outcome: Tearing
Description: Tearing will be reported according to the following scale: absent, mild, moderate and severe.
Time Frame: 10 days
Population: Intention-to-treat analysis (ITT)
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | PRO-155 Ophthalmic Solution 0.09 %
Number analyzed (Participants) | 35
Number analyzed (eyes) | 70
eyes
  right eye : absent | 34
  right eye : mild | 0
  right eye : moderate | 0
  right eye : severe | 0
  left eye : absent | 34
  left eye : mild | 0
  left eye : moderate | 0
  left eye : severe | 0
  left eye : Missing data | 1
  right eye : Missing data | 1

8. Secondary Outcome: Foreign Body Sensation
Description: Foreign body sensation will be reported according to the following scale: absent, mild, moderate and severe.
Time Frame: 10 days
Population: Intention-to-treat analysis (ITT)
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | PRO-155 Ophthalmic Solution 0.09 %
Number analyzed (Participants) | 35
Number analyzed (eyes) | 70
eyes
  right eye : absent | 34
  right eye : mild | 0
  right eye : moderate | 0
  right eye : severe | 0
  left eye : absent | 34
  left eye : mild | 0
  left eye : moderate | 0
  left eye : severe | 0
  left eye: Missing data | 1
  right eye : Missing data | 1

9. Secondary Outcome: Photophobia
Description: photophobia will be reported according to the following scale: absent, mild, moderate and severe.
Time Frame: 10 days
Population: Intention-to-treat analysis (ITT)
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | PRO-155 Ophthalmic Solution 0.09 %
Number analyzed (Participants) | 35
Number analyzed (eyes) | 70
eyes
  right eye : absent | 34
  right eye : mild | 0
  right eye : moderate | 0
  right eye : severe | 0
  left eye : absent | 34
  left eye : mild | 0
  left eye : moderate | 0
  left eye : severe | 0
  left eye : Missing data | 1
  right eye : Missing data | 1

10. Secondary Outcome: Chemosis
Description: chemosis will be reported according to the following scale: absent, mild, moderate and severe.
Time Frame: 10 days
Population: Intention-to-treat analysis (ITT)
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | PRO-155 Ophthalmic Solution 0.09 %
Number analyzed (Participants) | 35
Number analyzed (eyes) | 70
eyes
  right eye : absent | 34
  right eye : mild | 0
  right eye : moderate | 0
  right eye : severe | 0
  left eye : absent | 34
  left eye : mild | 0
  left eye : moderate | 0
  left eye : severe | 0
  left eye : Missing data | 1
  right eye : Missing data | 1

11. Secondary Outcome: Corneal Damage by Fluorescein Staining Test
Description: Corneal damage will be reported by Fluorescein eye staining using the following scale: absent, mild, moderate, and severe.
Time Frame: 10 days
Population: Intention-to-treat analysis (ITT)
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | PRO-155 Ophthalmic Solution 0.09 %
Number analyzed (Participants) | 35
Number analyzed (eyes) | 70
eyes
  right eye : absent | 34
  right eye : mild | 0
  right eye : moderate | 0
  right eye : severe | 0
  left eye : absent | 34
  left eye : mild | 0
  left eye : moderate | 0
  left eye : severe | 0
  left eye : Missing data | 1
  right eye : Missing data | 1

12. Secondary Outcome: Corneal Damage by Lissamine Green Staining Test
Description: Corneal damage will be reported by lissamine green staining using the following scale: absent, mild, moderate, and severe.
Time Frame: 10 days
Population: Intention-to-treat analysis (ITT)
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | PRO-155 Ophthalmic Solution 0.09 %
Number analyzed (Participants) | 35
Number analyzed (eyes) | 70
eyes
  right eye : absent | 34
  right eye : mild | 0
  right eye : moderate | 0
  right eye : severe | 0
  left eye : absent | 34
  left eye : mild | 0
  left eye : moderate | 0
  left eye : severe | 0
  left eye : Missing data | 1
  right eye : Missing data | 1

ADVERSE EVENTS:
Arm/Group | PRO-155 Ophthalmic Solution 0.09 %
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the information is confidential and exclusive property of the sponsor. Information can be revealed only to my staff and regulatory agencies or ethics committee.

All the information from this protocol is confidential and exclusive property of the sponsor, it can not be revealed without written consent from the sponsor.